CLINICAL TRIAL: NCT01848379
Title: Human Polymorphonuclear Neutrophil (PMN) Cytosolic Signaling and Effector Functions in Patients With Diabetes Mellitus Type 2 and Periodontitis
Brief Title: White Blood Cell Signaling and Defense Mechanisms in Patients With Diabetes Mellitus Type 2 and Periodontitis
Acronym: DMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zentrum fuer Zahn-, Mund- und Kieferheilkunde (Other)
Responsible Party: Principal Investigator, Dr. Jens Martin Herrmann, research associate, Zentrum fuer Zahn-, Mund- und Kieferheilkunde
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DMS017507GI
Record Dates: First submitted 2013-04-29; First posted 2013-05-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Chronic Periodontitis; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Antidiabetic Therapy(ADT)+Full Mouth Decontamination(FD) (Experimental): ADT:
  (Par-)enteral, anti-diabetic medication, diet and dietetic supervision, physiotherapy and physical exercises
  FD:
  The oral use of topical antiseptics prior and after mechanical tooth debridement, tooth as well as root surface planing and soft tissue decontamination in combination with systemic antibiotics (a combination of amoxicillin and metronidazole - if no microbial resistances were detected)
  Interventions: Procedure: ADT+FD
- Full Mouth Deconatamination(FD) (Active Comparator): FD:
  The oral use of topical antiseptics prior and after mechanical tooth debridement, tooth as well as root surface planing and soft tissue decontamination in combination with systemic antibiotics (a combination of amoxicillin and metronidazole - if no microbial resistances were detected)
  Interventions: Procedure: FD
- No Treatment (No Intervention): Healthy individuals to be monitored cross-sectional

INTERVENTIONS:
Procedure: ADT+FD
  Other Names: Anti-diabetic Treatment and Full Mouth Decontamination
  Arms: Antidiabetic Therapy(ADT)+Full Mouth Decontamination(FD)
Procedure: FD
  Other Names: Full Mouth Decontamination
  Arms: Full Mouth Deconatamination(FD)

SUMMARY:
White blood cell membrane and surface structures are affected by the metabolic disorders and complications found in diabetes mellitus. Therefore, cellular activation, signal propagation, intracellular signaling as well as bactericidal effector functions are altered.

When diabetic symptoms are corrected by the systemic intervention and treatment of the patients (Anti-diabetic Therapy/ADT, i.e. anti-diabetic medication, diet and dietetic supervision, physiotherapy and physical exercises), white blood cell functions will then normalize and reach the functionality comparable to those cells derived from healthy subjects.

Gum diseases like periodontitis have long been associated with and termed complications of uncontrolled diabetes mellitus. Vice versa, after diabetic conditions are corrected, periodontitis treatment will be proven effective, when oral hygiene regimen, full mouth decontamination (FD, i.e. the oral use of topical antiseptics prior and after professional mechanical tooth cleaning, tooth as well as root surface planing, polishing as well as gum and soft tissue decontamination in combination with systemic antibiotics) are performed. To reinforce gum healing, reinfection prevention (RP) as well as supportive periodontal therapy (SPT) will be administered by dental professionals on an individual basis and a detailed schedule.

If periodontal pockets critical for participant's self care are not eliminated by FD including RP and SPT, and niches >5mm after 6 month persist, patients are informed and offered surgical intervention as indicated for gum disease elimination.

Dental follow up exams will be offered to all participants.

DETAILED DESCRIPTION:
Specific Aims

1. To investigate if cytosolic Ca2+- ( delta[Ca2+]i) and pH (delta_pHi) signaling responses and bactericidal effector functions of PMN dependent upon the status of diabetic control and are reduced or increased when compared to age and gender matched controls
2. To determine the biochemical basis for diabetic PMN alteration of motility as well as bactericidal functions: production of superoxide and release of elastase, respectively
3. To characterize the molecular basis of the observed alterations in the regulation of cytosolic calcium (delta[Ca2+]i) and pH (delta_pHi) exhibited by diabetic PMN
4. To investigate if the pre-activated state and altered bactericidal functionality of diabetic PMN are reversed when the patients' glycemic control is normalized, blood glucose levels as well as periodontal disease are corrected
5. To evaluate, if systemic and periodontal intervention can lead to clinical attachment gain in patients with diabetes mellitus type 2

ELIGIBILITY:
Inclusion Criteria:

* Diabetes Mellitus, Type II
* Glycated Hemoglobin ≥8.5%
* Chronic Periodontitis
* Patients and controls should have at least 12 natural teeth (without subgingival fillings, crowns or caries)

Exclusion Criteria:

* Pregnancy
* Smoking
* Low Body Mass Index (BMI <18.5kg/m*m)
* Severe cardiovascular disease including coronary artery disease, cerebral vascular disease, peripheral vascular disease, valvular heart disease, and congestive heart failure
* Other major illnesses including cancer, liver disease, pulmonary disease, chronic infectious disease other than periodontitis (HIV, hepatitis, etc.), rheumatological disease, hematological disease, or any condition requiring hospitalization or chronic medical therapy other than diabetes.
* Major psychiatric illness requiring treatment, or that might interfere with the ability to understand or cooperate with the protocol
* Ongoing alcohol or drug abuse; all forms of medication or illegal substance abuse
* Systemic enteral or parenteral medication, in part daily vitamin or anti-oxidative supplementation and certain calcium channel blockers (i.e. Nifedipine); but anti diabetic drugs or insulin substitution
* Allergies to antibiotics or adjuvant medication / antiseptics as well as dental materials in use (including gloves) in particular those against topical antiseptic solutions i.e. chlorhexidine / N',N'''''-hexane-1,6-diylbis[N-(4-chlorophenyl)(imidodicarbonimidic diamide)] or povidone iodine / 2-Pyrrolidinone, 1-ethenyl-, homopolymer, compound with iodine
* Severe dental disease defined as severe dental caries, and/or severe pulpal disease requiring surgical correction, or any other mucosal or dental condition not readily treated, or requiring extensive dental, oral surgical or prosthetic treatment, or any other oral treatment which could affect the outcome of periodontal therapy or diseases or syndromes that require systemic medication.
* Systemic, topical or inhaled steroid treatment for more than 30 consecutive days within 6 weeks of baseline.
* Any periodontal treatment within 6 months prior to baseline
* For controls: a periodontal screening index (PSI) > 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Clinical Attachment Level (CAL) at 6 and 12 Months | 0, 6 and 12 months
  CAL: Clinically and quantitatively, level of attachment is defined as the distance in mm from the cemento-enamel junction (CEJ) of the teeth to the bases of the periodontal pockets. Attachment gain may be found during healing or periodontal treatment procedures.

SECONDARY OUTCOMES:
Probing Pocket Depth (PPD) | 0, 6 and 12 months
  PPD: also called periodontal probing depth is defined as the distance in millimeters from the gingival margin to the base of the sulcus or periodontal pocket. It is measured on six surfaces/tooth (disto-buccal, mid-buccal, mesio-buccal, disto-lingual, mid-lingual, and mesio-lingual) of all teeth present using the pressure calibrated Florida probe.
Bleeding on Probing (BOP) | 0, 6 and 12 months
  BOP: will be determined by recording the presence or absence of bleeding following probing to determine pocket depth (PPD). This parameter will be expressed as % bleeding sites out of all examined sites in the dentition and will be documented with the Florida probe software.
Body Mass Index (BMI) | -3 weeks; 0, 6 and 12 months
  The body mass index will be assessed as the participants' body mass divided by the square of their height
Glycated Hemoglobin (HbA1c) | -3 weeks; 0, 6 and 12 months
  Physiological levels of blood glucose result in a normal amount of glycated hemoglobin. Treatment procedures may help to reduce plasma glucose in individuals with diabetes mellitus type 2, thus, in a timely extended fashion the fraction of glycated hemoglobin.

OTHER OUTCOMES:
Neutrophil Cytoplasmic Calcium Concentration ([Ca2+]i) | -3, 0 and 2 weeks; 6 and 12 months
  [Ca2+]i: ex vivo 2nd messenger cytoplasmic calcium concentration resembles a key parameter for chemoattractive or phagocytic PMN-receptor activation.
Neutrophil Cytoplasmic pH (pHi) | -3, 0 and 2 weeks; 6 and 12 months
  pHi: ex vivo liganded neutrophil receptors initiate a series of signals, resulting in phagocytosis of an entity and release of the phagocyte granules' contents as well as oxidative products. The specific mechanisms by which these effector functions occur depend upon the receptor involved among [Ca2+]i is changes of pHi.
Release of Reactive Oxygen Species (ROS) | -3, 0 and 2 weeks; 6 and 12 months
  ROS: these NADPH products are predominantly found within phagolysosomal compartments of the neutrophils. During phagocytosis, neutrophils may release ROS resulting in collateral tissue damage. The reactivity of ROS release will be assessed ex vivo after activation of chemoattractant as well as phagocytic receptors of the cells.
Release of Neutrophil Elastase (EA) | -3, 0 and 2 weeks; 6 and 12 months
  EA: residing in the azurophilic granules of the neutrophils, elastase is activated after phagolysosomal fusion; thence, in proximity to the engulfed entities it unfolds bactericidal activity by degrading valine-rich proteins. The elastolytic activity will be assessed ex vivo after chemoattractant as well as phagocytic activation of the neutrophils' receptors.
Gingival Crevicular Fluid (GCF) | -3 and 0 weeks
  GCF: a quantitative and qualitative assessment of the serum like exudate in the gingival crevice will be performed.
Global Luminol Dependent Chemiluminescence of Stimulated Neutrophils (CLt) | 0 weeks
  The detection of total ROS will be performed ex vivo with a kinetic chemiluminescence assay after receptor activation of neutrophils.
Extracellular Luminol Dependent Chemiluminescence of Stimulated Neutrophils (CLex) | 0 weeks
  The detection of extracellular ROS will be performed ex vivo with a kinetic chemiluminescence assay after receptor activation of neutrophils.
Cellular Immune responses | 0, 6 and 12 months
  Analyses of leukocyte subsets, i.e. T-lymphocytes from the peripheral venous blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Jens Martin Herrmann, Dr., Principal Investigator — Department of Periodontology, ZentrumZMK
Locations (1):
- Department of Periodontontology, ZentrumZMK, Giessen, Germany

REFERENCES:
- [Derived] Herrmann JM, Sonnenschein SK, Groeger SE, Ewald N, Arneth B, Meyle J. Refractory neutrophil activation in type 2 diabetics with chronic periodontitis. J Periodontal Res. 2020 Apr;55(2):315-323. doi: 10.1111/jre.12717. Epub 2020 Jan 8. PMID 31912903